CLINICAL TRIAL: NCT04229173
Title: Natural History and Disease Progression Biomarkers of Multiple System Atrophy
Acronym: ASPIRE-MSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/19/0161
Record Dates: First submitted 2019-11-28; First posted 2020-01-18 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Multiple System Atrophy
Keywords: MSA; MRI; Dat spect; Atrophy; Biomarkers
MeSH Terms: conditions — Multiple System Atrophy; Atrophy | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSA patients (Other): Patients with multiple system atrophy will be examined at baseline, 6 months and 12 months via the following procedures performed at all 3 visits:
  * a clinical examination;
  * blood and cerebrospinal fluid (CSF) (optional) sampling for the assessment of selected fluid biomarkers;
  * MRI for the assessment of brain volume, white matter integrity and cerebral iron deposition; DAT-SPECT (Dopamine Transporter, Single Photon Emission Computed Tomography) for the assessment of presynaptic dopaminergic function
  Interventions: Diagnostic Test: MRI acquisition; Diagnostic Test: DAT-SPECT; Diagnostic Test: blood sample, cerebrospinal fluid (optional); Behavioral: Evaluations about motor abilities, depression, cognition and lifestyle
- Healthy volunteers (Other): healthy. Controls will undergo an MRI scan at baseline, 6 months and 12 months, and a DAT-SPECT(Dopamine Transporter, Single Photon Emission Computed Tomography) scan at baseline and 12 months.
  Interventions: Diagnostic Test: MRI acquisition; Behavioral: Evaluation about depression cognition

INTERVENTIONS:
Diagnostic Test: MRI acquisition — MRI acquisition
Diagnostic Test: DAT-SPECT — Imaging with DAT SPECT (Dopamine Transporter, Single Photon Emission Computed Tomography)
  Arms: MSA patients
Diagnostic Test: blood sample, cerebrospinal fluid (optional) — blood sample, cerebrospinal fluid
  Arms: MSA patients
Behavioral: Evaluations about motor abilities, depression, cognition and lifestyle — Evaluations about motor abilities (UMSAR scale), depression (BDI scale), cognition (MoCA scale) and lifestyle (MSA- QoL)
  Arms: MSA patients
Behavioral: Evaluation about depression cognition — Evaluations about depression (BDI scale), cognition (MoCA scale)
  Arms: Healthy volunteers

SUMMARY:
Multiple system atrophy (MSA) is a rare and fatal neurodegenerative disease characterised by a variable combination of parkinsonism, cerebellar impairment and autonomic dysfunction. The neuropathological hallmark is the accumulation of alpha-synuclein in oligodendrocytes. While some symptomatic treatments exist, neuroprotective treatments for MSA remain an urgent, unmet need. Moreover, at present there is not a single surrogate biomarker of MSA which could be used to inform clinical trials.

This study seeks to characterise the natural history of MSA on a panel of candidate biomarkers, pre-selected for being putative surrogates of the underlying neurodegenerative process

DETAILED DESCRIPTION:
Surrogate biomarkers are objectively measured characteristics of a disease which act as indicators of the underlying pathophysiological processes responsible for disease progression. Reduced grey matter volume in putamen, cerebellum and brainstem as measured with MRI have been consistently reported to differentiate MSA from other parkinsonian disorders. However, to date, there are no longitudinal studies examining the natural history of MSA on these structural neuroimaging markers over time. The magnitude of the abnormalities observed cross-sectionally in MSA compared to other parkinsonian disorders and the fast clinical progression of the disease make it very likely that structural changes can be observed even over short periods of time. There is also a strong scientific rationale for the potential of measures reflecting white matter integrity, cerebral iron deposition and presynaptic dopaminergic dysfunction, as well as levels of neurofilament light chain (NfL), alpha-synuclein and other proteins involved in the neurodegenerative process in MSA, to serve as progression biomarkers of the disease, although supporting evidence remains limited. A better understanding of the natural history of MSA over 6 and 12 months on a panel of candidate surrogate biomarkers is needed to better understand the disease, help optimise future trial designs in terms of patient selection, sample size and trial duration, and improve the ability to measure the therapeutic effects of novel treatments.

In evaluating potential progression markers of a neurodegenerative disease such as MSA, it is important to control for the normal effects of aging. Studies in healthy volunteers have shown regionally distinct effects of aging on both brain volume and dopamine transporter density, justifying the inclusion of healthy controls with a similar age and gender distribution than patients.

ELIGIBILITY:
INCLUSION CRITERIA:

Applicable to MSA patients:

* Patients with possible or probable MSA according to consensus diagnosis criteria [Gilman et al., 2008]
* Patients aged between 30 and 80 years
* Patients at the early stages of the disease, defined as maximum 5 years since the onset of one of the following symptoms associated to MSA:

Parkinsonism Ataxia Orthostatic hypotension and/or urinary dysfunction - Patients with an anticipated survival of at least 3 years on the basis of Investigators' clinical judgment

Applicable to healthy controls:

* Participants with a similar age (+/- 5 years) and gender distribution compared to MSA patients
* Participants with absence of neurological pathology
* Patients aged between 25 and < 80 years

Applicable to both patients and healthy controls:

- Participants who voluntarily sign the written informed consent form, indicating that they understand the purpose of and procedures required for the study and are willing to participate in it Participants affiliated to the French social security health system

EXCLUSION CRITERIA:

Applicable to MSA patients:

* Speech impairment (score of ≥3 on UMSARS (Unified Multiple System Atrophy Rating Scale) question 1);
* Impairment in ambulation (score of ≥3 on UMSARS (Unified Multiple System Atrophy Rating Scale) question 7)
* Falling more frequently than once per week (score of ≥3 on UMSARS (Unified Multiple System Atrophy Rating Scale) question 8)

Applicable to both MSA patients and healthy controls:

* Participants with significant cognitive impairment (MoCA score <21)
* Any major medical or psychiatric condition which may compromise participation in the study or the safety, at the discretion of the Investigator
* Contraindications for MRI imaging, including claustrophobia and presence of metallic implants such as cardiac or auditory prostheses, pacemakers or cerebral clips
* Contraindications to obtain a FP-CIT SPECT(Single Photon Emission Computed Tomography) (i.e. known hypersensitivity to the active substance or to any of the excipients, or to iodine)
* Current pharmacological treatments that may alter the DAT(dopamine transporter ) SPECT (Single Photon Emission Computed Tomography) reading, including amphetamines, benzatropine, buproprion (amfebutamone), cocaine, mazindol, methylphenidate, phentermine or sertraline
* Females who are pregnant, breast feeding or of child bearing age without effective contraception
* Participants who lack the capacity to give informed consent
* Participants taking any investigational products within 3 months before baseline assessment
* Participant under adult autonomy protection system, legal guardianship or incapacitation.

Additional exclusion criteria concerning only patients consenting to the lumbar puncture:

* Coagulopathy and/or anticoagulant treatment
* Thrombocytopenia
* Intracranial hypertension
* Severe degenerative arthritis of the lumbar spine Patients failing to meet these criteria can still participate in the study and all other study assessments (with the exception of lumbar puncture) as appropriate.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Change putamen, cerebellum and brainstem volume measured on MRI | at 12 month
  volume measured with T1-3D MRI, unit : Volume (mm3), Fer: R2* (s-1), diffusion: mean diffusivity (mm2s-1)

SECONDARY OUTCOMES:
Effect of disease progression on other measures of brain structural integrity and iron accumulation | 6 month and 12 month
  volume measured with T1-3D MRI, unit : Volume (mm3), Fer: R2* (s-1), diffusion: mean diffusivity (mm2s-1)
Effect of disease progression on the loss of presynaptic dopaminergic terminals in the striatum integrity and iron accumulation | 6 month and 12 month
  volume measured with DAT SPECT (Single Photon Emission Computed Tomography), unit : binding potential (e.g ratio striatum/brain activity)
Effect of disease progression on axonal damage as evidenced in biofluids | 6 month and 12 month
  biomarkers dosages in blood and Cerebral Spinal Fluid total Concentration unit : pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier RASCOL, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (10):
- France (10):
  - CHU de Bordeaux, Bordeaux
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - Chu Clermont Ferrand, Clermont-Ferrand
  - CHU Lille, Lille
  - Hôpital de La Timone, Marseille
  - CHU de Nancy, Nancy
  - Clinique neurologique - Hôpital Laennec, Nantes
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital de Hautepierre, Strasbourg
  - CHU, Toulouse